CLINICAL TRIAL: NCT03249441
Title: Compassion-Focused Therapy for People With Severe Obesity: A Randomised Controlled Study.
Brief Title: Compassion-Focused Therapy for People With Severe Obesity.
Acronym: CFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Mary Hynes, Mary Hynes, Senior Clinical Psychologist, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUIreland
Record Dates: First submitted 2017-07-31; First posted 2017-08-15 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: This study utilised a randomised controlled trial (RCT) research design to investigate the efficacy of a group based CFT intervention programme. Participants were randomly allocated to one of the two groups, CFT plus Treatment as Usual (CFT) or Treatment As Usual (TAU), and psychological measures were administered at three time points (pre-intervention, post-intervention and follow-up assessment at three months follow up). The primary outcomes included self-compassion, shame and self-criticism. Emotional eating and depressive symptoms were assessed as secondary outcomes.
Who Masked: Outcomes Assessor
Masking Description: Clients are randomly assigned to one of two groups, Treatment as Usual (TAU) or Compassion-focused therapy plus Treatment as Usual (CFT). The outcomes assessor is blind to which of the two groups participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compassion-focused therapy (Experimental): Compassion-Focused Therapy (CFT) Participants were taught the main compassion-focused exercises as outlined in 'The Compassion-Mind Guide to Ending Overeating: Using Compassion-Focused Therapy to overcome Bingeing and Disordered Eating' manual (Goss, 2011) over a ten session period (weekly for 2 hours), offered over a 3 month period. Self-criticism and shame were key foci across sessions. Participants in the CFT arm also received Treatment as Usual.
  Interventions: Behavioral: Compassion-focused therapy
- Treatment as Usual (No Intervention): Treatment As Usual Treatment as usual was based in the Diabetes, Endocrinology and Metabolism Clinic in Galway University Hospital. The Weight Management Service provides assessment by a multi-disciplinary team of endocrinologists, dieticians, nurse specialists and clinical psychologists. Dietary advice is given by a specialist dietician regarding weight management, assessment by the Consultant Endocrinologist with possible medication for management of diabetes and weight, and participation in a healthy lifestyle education program.

INTERVENTIONS:
Behavioral: Compassion-focused therapy — Session-by-session summary of CFT:
  Week 1: Understanding your relationship with food Week 2: Making sense of overeating Week 3: The Compassionate Mind/ Preparing your mind for compassion Week 4: Developing the skill of self-compassion Week 5: Why we overeat - a Compassionate approach Week 6: Understanding your current eating pattern Week 7: Motivating yourself to change Week 8: Determining what your body needs Week 9: Towards a new way of eating Week 10: Compassionate letter writing and developing a compassionate focus on eating.
  __________________________________________________________________________
  Arms: Compassion-focused therapy

SUMMARY:
This study aims to explore the effectiveness of a group psychotherapy intervention using Compassion-Focused Therapy (CFT) in adults with severe obesity. In particular, it aims to evaluate the principle that CFT can be used to reduce levels of shame and self-criticism in adults with severe obesity

OBJECTIVES:

The objective of the current study is to assess and compare a CFT group intervention to Treatment as Usual (TAU) with regard to psychological functioning, specifically self-compassion, shame, self-criticism, emotional eating and mood.

DETAILED DESCRIPTION:
Compassion-focused therapy (CFT) was specifically designed for people with high levels of shame, self-criticism and self-directed hostility by helping people to cultivate affiliative emotions and compassion.The current research aims to explore changes in levels of self-criticism, shame, submissive behaviour, and self-comparison in a severely obese population who are awaiting bariatric surgery. As depression symptoms and levels of emotional eating can interfere with bariatric surgery success, these constructs are included as secondary outcomes for research.

Research questions

The research was guided by the following research questions and hypotheses:

1. Does CFT significantly improve levels of self-compassion and social comparison?

   Hypotheses:
   1. It was hypothesised that CFT would show significant improvements in comparison to TAU on self-compassion and social comparison variables.
   2. It was hypothesised that these improvements would be maintained at 3 months follow up.
2. Is CFT effective in reducing levels of shame, self-criticism and submissive behaviour for people who are severely obese?

   Hypotheses:
   1. It was hypothesised that CFT would achieve significant reductions in shame, self-criticism, and submissive behaviour variables in comparison to TAU.
   2. It was hypothesised that these changes would be maintained at 3 months follow up.
3. Does CFT reduce emotional eating and depression?

Hypotheses:

1. It was hypothesised that CFT would show significant reductions in emotional eating and depression variables in comparison to TAU.
2. It was hypothesised that these reductions would be maintained at 3 months follow up.

This study will use a prospective, randomised control design using quantitative methods to investigate the effectiveness of CFT, using various measures pre-and post-therapy and at 3-month follow-up.

91 individuals with severe obesity will be randomly assigned to one of two treatment groups

- Compassion-Focused Therapy (CFT) plus treatment as usual or Treatment as Usual alone (TAU).

Individuals assigned to CFT will be introduced to the CFT model taught the main compassion-focused exercises in a group setting. Self-report measures will be administered prior to the commencement of the CFT group and TAU group, and during the final groups and 3 months follow up. To reduce the 'demand' effect, scales will be administered by an Assistant Psychologist who is not involved in delivering the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a clinical diagnosis of Severe Obesity, as defined by a Body Mass Index (BMI) of 40 kg/m² or more
* Participant is aged 18 years or older
* Participant is not in receipt of psychological interventions at the time of randomisation to group

Exclusion Criteria:

* Participant has insufficient English language ability to take part in the group and complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
Self-compassion | 6 months
  The Self-Compassion Scale, Short Form (SCS-SF). This is a 12-item self-report measure, developed by Neff (2003).

SECONDARY OUTCOMES:
Shame | 6 months
  Shame (the Other as Shamer Scale;OAS) The OAS is an 18- item scale developed by Goss, Gilbert, and Allan (1994).Participants respond to statements such as 'I think that other people look down on me' on a five-point Likert scale according to the frequency with which they make certain evaluations about how others judge them (0 = never, to 5 = almost always).
Self-criticism | 6 months
  The Forms of the Self-Criticising/Attacking and Self-Reassuring Scale (FSCRS). This scale was developed by Gilbert, Clark, Hempel, Miles, and Irons (2004). It was developed to measure self-criticism and the ability to self-reassure.
Submissive Behaviour | 6 months
  Submissive Behaviour Scale (SBS). This scale was originally developed from the work of Buss and Craik (1986). The most highly agreed upon items were chosen to construct the Submissive Behaviour Scale (Allan & Gilbert, 1997).
Social Comparison | 6 months
  Social Comparison Scale (SCS). This scale was developed by Allan and Gilbert (1995) to measure self-perceptions of social rank and relative social standing

OTHER OUTCOMES:
Mood | 6 months
  Beck Depression Inventory-II (BDII; Beck, Steer, & Brown, 1996). The BDI-II is a widely used, 21-item self-report measure of depressive symptomatology which requires participants to respond to statements describing symptoms of depression on a scale rated 0 (never) to 3 (always).
Emotional Eating | 6 months
  The Emotional Eating Scale (EES). This scale measures the use of eating to cope with negative mood. Responders are asked to rate the strength of their urge to eat (in one of five categories ranging from 'no urge to eat' to 'overwhelming urge to eat') in relation to 25 different emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Hynes, M.Psych.Sc, Principal Investigator — National Univeristy of Ireland, Galway

IPD SHARING:
Plan to Share IPD: No